CLINICAL TRIAL: NCT06973070
Title: Utilization of Upper GI Marshmallow Series Versus High Resolution Manometry in Preoperative Esophageal Motility Assessment
Brief Title: Upper GI MM vs Manometry
Status: Completed | Type: Observational
Sponsor: Lexington Health Incorporated (Other)
Responsible Party: Principal Investigator, Marc Antonetti, MD, Principal Investigator, Lexington Health Incorporated
Other Study IDs: LMCII2025-003
Record Dates: First submitted 2025-05-05; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-03

CONDITIONS: GERD (Gastroesophageal Reflux Disease)
Keywords: GERD REFLUX GASTRIC REFLUX
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Research will consist of retrospective review of prospective cohort quantitative data collection with the goal of comparing preoperative High-Resolution Manometry (HRM) results to Upper Gastrointestinal Marshmallow (UGIMM) results, in the patient undergoing preoperative esophageal motility assessment. The aim of this study is to establish a correlation between HRM and UGIMM studies in order to create a clinically supported gold standard measurement for preoperative esophageal motility assessment. Research will examine the level of reliability and variability of the esophageal motility assessment conducted utilizing HRM and the UGIMM study. Standards of testing and current practice guidelines will be reviewed and compared for correlations in procedure outcomes. Research seeks to accomplish validation and strengthening of current practices related to the use and interpretation of HRM and UGIMM study results as a valid postoperative outcome predictor.

DETAILED DESCRIPTION:
Identifying esophageal motility disorders prior to surgical intervention is imperative when determining the procedural route that will produce the greatest positive patient outcome and reduce postoperative sequelae related to preoperative conditions. Possible disparities have been identified between HRM and UGIMM assessment results. Identifying testing variables and standards that could impact the obtained results will allow providers the ability to create a more customized plan of care and increase outcome predictability. Therefore, examining HRM and UGIMM level of agreement is essential to providing the best evidence-based practice care and meeting the unique needs of individual patients.

Currently, HRM results are noted as the standard benchmark for adequate assessment of esophageal motility function and disorders. Esophageal manometry testing provides a means to determine if the esophagus is functioning properly through a series of wet swallows. As a patient swallows, the esophagus contracts in an orderly sequence to push the swallowed contents into the stomach. Once the contents enter the stomach, the Lower Esophageal Sphincter (LES) closes to prevent backflow, or reflux, of stomach contents into the esophagus. Any impairment to esophageal motility can compromise clearance and sphincter function, leading to adverse outcomes such as the development of intestinal metaplasia due to prolonged exposure of the mucosa to gastric acid. Assessment of motility and sphincter function is vital prior to any surgical intervention that involves manipulation of the gastroesophageal junction (GEJ) or surrounding structures. Inaccurate surgical manipulation can cause undesired pressure changes and alterations in normal peristalsis within the esophageal body.

By assessing preoperative baseline esophageal function, postoperative changes can be better predicted and adequacy of surgical intervention assessed. Some studies have noted that HRM metrics can predict overall surgical response and postoperative outcomes. Identification of motility dysfunction, or an incompetent LES, can be obtained during this examination, even in asymptomatic patients.

During HRM testing a flexible, small-bore probe will be passed via the nasal passages, down the esophagus and into the stomach. The patient is then asked to swallow a 5-milliliter saline fluid bolus while in the supine position for an average of 10 swallows. The test is then repeated in the standing, or upright, position for comparison. Pressure sensors on the probe record esophageal pressure, motility configurations, and contraction patterns. During the examination data is transmitted, via the probe, to a software program with the capability to autogenerate an analysis and diagnosis of the data. However, the autogenerated analysis can be situationally limited, therefore, the test administrator must possess a high level of understanding and keen interpretation skills to produce a completely accurate diagnosis. During study analysis it is often necessary to adjust anatomical markers, such as the location of the LES, Upper Esophageal Sphincter (UES), and the diaphragm, as the preset software data is unable to compensate for certain situational factors that may impact marker placement, such as GEJ morphology. The test administrator will identify and mark the UES, LES, and the pressure inversion point (PIP) during the interpretation phase. The integrated relaxation pressure (IRP) is then autocalculated, and provides a measurement of deglutitive relaxation during a 10 second time frame after the swallow is completed. The distal contractile integral (DCI) is also auto calculated and measures dynamism of peristalsis within the muscles of the esophagus. The PIP allows for evaluation of transition from the intra-abdominal cavity to the intrathoracic cavity. HRM results are categorized using the standardized Chicago Classification system which is subdivided into 4 hierarchical categories: 1) incomplete LES relaxation, 2) major motility disorders, 3) minor motility disorders, and 4) normal esophageal motility. Given that the test administrator has the ability to manipulate measurement markers during the analysis process, the need exists to identify possible gaps in consistency among test administrators, examine expected HRM results against other testing measures, such as the UGI MM test, and determine the impact the results have on patient outcomes.

A less invasive alternative to the HRM test is the UGIMM study. The UGIMM study is conducted under fluoroscopy and allows for the evaluation of motility function in real time, as well as visualization of anatomical structures. During the procedure radiographs are taken while the patient swallows a self-defined sip of barium in the standing position. The patient is then placed in the Trendelenburg position and asked to swallow a barium-soaked marshmallow while another set of radiographic images are taken. Each marshmallow measures the same, weighing approximately 6 grams. The UGIMM study currently does not have an established classification system by which result measurements are validated. However, exam outcomes are generally measured as follows: normal if the bolus clears the esophagus within 2 swallows or less; borderline swallowing dysfunction if the bolus clears within 3-4 swallows; abnormal swallowing function if 5 or more swallows are required to clear, or if a portion of the bolus remains after 5 swallows.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative patients who have undergone both HRM and UGIMM assessments as part of their preoperative plan of care.
2. Patients who have had surgical procedures involving the upper GI tract and immediate surrounding structures after completing HRM and UGIMM assessments preoperatively.
3. Adults aged 18 and older.

Exclusion Criteria:

1. Patients who continued taking narcotics, calcium channel blockers, nitrates, or promotility medications the day of the HRM test, as these medications could falsely relax or hyper stimulate esophageal structures (Snyder & Ravi, 2021).
2. Patients with a past surgical history that includes Heller myotomy, peroral esophageal myotomy, botulinum injections, pneumatic dilations, or gastric fundoplication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing preoperative testing for surgical intervention involving manipulation of the upper gastrointestinal tract.
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
The aim of this study is to establish a correlation between High Resolution Manometry and Upper Gastrointestinal Marshmallow studies to create a clinically supported gold standard measurement for preoperative esophageal motility assessment | September 2020-April 2024
  Research will examine the level of reliability and variability of the esophageal motility assessment conducted utilizing High Resolution Manometry and the Upper Gastrointestinal Marshmallow study. Standards of testing and current practice guidelines will be reviewed and compared for correlations in procedure outcomes. Research seeks to accomplish validation and strengthening of current practices related to the use and interpretation of High Resolution Manometry and Upper Gastrointestinal Marshmallow study results as a valid postoperative outcome predictor.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Antonetti, MD, Principal Investigator — Lexington Health Incorporated
Locations (1):
- Lexington Health Incorporated, West Columbia, South Carolina, United States

REFERENCES:
- [Background] Musella M, Vitiello A, Berardi G, Velotti N, Pesce M, Sarnelli G. Evaluation of reflux following sleeve gastrectomy and one anastomosis gastric bypass: 1-year results from a randomized open-label controlled trial. Surg Endosc. 2021 Dec;35(12):6777-6785. doi: 10.1007/s00464-020-08182-3. Epub 2020 Dec 2. PMID 33269429
- [Background] FalcAo AM, Nasi A, Szachnowicz S, Santa-Cruz F, Seguro FCBC, Sena BF, Duarte A, Sallum RA, Cecconello I. Does the nissen fundoplication procedure improve esophageal dysmotility in patients with barrett's esophagus? Rev Col Bras Cir. 2020 Nov 30;47:e20202637. doi: 10.1590/0100-6991e-20202637. eCollection 2020. English, Portuguese. PMID 33263652
- [Background] Yadlapati R. High-resolution esophageal manometry: interpretation in clinical practice. Curr Opin Gastroenterol. 2017 Jul;33(4):301-309. doi: 10.1097/MOG.0000000000000369. PMID 28426462
- See also: Related Info — http://www.ncbi.nlm.nih.gov/books/NBK559237